CLINICAL TRIAL: NCT06087731
Title: Efficacy and Safety of Tocilizumab for Patients With Thyroid-associated Ophthalmopathy
Brief Title: Efficacy and Safety of Tocilizumab for TAO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: For some personal reasons.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, Dan Liang, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023TAOIL-6
Record Dates: First submitted 2023-09-22; First posted 2023-10-18 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-04

CONDITIONS: Tocilizumab; Thyroid Associated Ophthalmopathy
Keywords: Thyroid Associated Ophthalmopathy; tocilizumab
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tocilizumab (Experimental): administrated with tocilizumab (8mg/kg) every four weeks
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab (8mg/kg) every 4 wekks

SUMMARY:
This study aims to evaluate the efficacy and safety of tocilizumab treating Thyroid Associated Ophthalmopathy.

DETAILED DESCRIPTION:
Thyroid Associated Ophthalmopathy(TAO) is one of autoimmune orbital diseases characterized by enlargement of the extraocular muscles and increase in fatty or/and orbit connective tissue volume affecting the appearance and visual function of the eyes. In TAO pathogenesis, orbital fibroblasts are activated by autoantibodies against the thyrotropin receptor TSHR and the insulin-like growth factor-1 receptor. The fibroblasts then secrete interleukin-6 (IL-6), macrophage chemoattractant protein-1, and transforming growth factor-ß. In orbital preadipocyte fibroblasts, IL-6 increases expression of the thyrotropin receptor TSHR, and the orbital volume is relative to IL-6 mRNA expression. Thus, IL-6 may have several roles in the pathogenesis of TAO. Tocilizumab, a recombinant humanized IgG1 monoclonal antibody against IL-6 receptors, is FDA-approved for the treatment of rheumatoid arthritis, giant cell arteritis and juvenile idiopathic arthritis with a good toleration. The investigators carry this perspective cohort study to evaluate the efficacy of tocilizumab in TAO.

ELIGIBILITY:
Inclusion criteria:

Age 18-70 years old

* Clinical diagnosis of Thyroid-associated ophthalmopathy
* Euthyroid status at least 1 months before baseline.
* No previous specific therapy for TAO, except for local measures
* Written informed consent is obtained

Exclusion criteria:

* Uncontrolled diabetes or hypertension
* Renal or hepatic insufficiency.
* Infectious diseases (HIV, HBV,TB and so on)
* History of mental/psychiatric disorder
* Other ocular diseases or fundus diseases.
* Any previous systemic medications or surgery for the treatment of TAO
* Pregnant or lactating females.
* Intolerability of tocilizumab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-23 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
volume and signal intensity of each extraocular muscles and soft tissue in MRI images | month 1，month 3，month 6
  The volume and signal intensity of each extraocular muscles and soft tissue are analyzed in the MRI slides of each patients. each part of each extraocular muscles and soft tissue were measured three times and two trained performers will do this assignment respectively.
Clinical Activity Score | month 1，month 3，month 6
  Spontaneous orbital pain. Gaze evoked orbital pain. Eyelid swelling that is considered to be due to active (inflammatory phase) GO. Eyelid erythema. Conjunctival redness that is considered to be due to active (inflammatory phase) GO (ignore "equivocal" redness).
  Chemosis. Inflammation of caruncle or plica
eyelid aperture | month 1，month 3，month 6
  For the assessment of eyelid aperture, the same millimeter ruler should be used by the same observer. When performed this assessment, participants should relax their eyes and keep looking ahead and the observers should keep the ruler perpendicular to their eyelid.
exophthalmos | month 1，month 3，month 6
  For the assessment of exophthalmos, the same Hertel instrument and ideally the same observer should be used on each occasion. Additionally the same intercanthal distance (ICD) should be used on each occasion.
eyelid lag | month 1，month 3，month 6
  For the assessment of eyelid aperture, the same millimeter ruler should be used by the same observer. Lid lag is defined that the lid margin distance in downgaze. The upper eyelid positions above (recorded '+') or below (recorded '-') the superior limbus will be measured in millimeters.
retraction of the upper and lower eyelids | month 1，month 3，month 6
  For the assessment of eyelid aperture, the same millimeter ruler should be used by the same observer. The upper eyelid positions above (recorded '+') or below (recorded '-') the superior limbus and the lower eyelid positions above (recorded '+') or below (recorded '-') the posterior limbus will be measured in millimeters on the primary position with relaxed status.

SECONDARY OUTCOMES:
ocular motility | month 1，month 3，month 6
  The head of each participant is adjusted to fix on the modified perimeter and set the visual axis of the examined eye on the center of the optimal visual target in visual chart. The other eye should be covered. The participantshould move the examined eye to follow the movement of the visual target until he/she cannot identify the exact visual target in vertical and horizontall directions respectively. And the extreme scales of these four directions (upgaze, downgaze, abduction and adduction) for each eye are obtained.
Graves' Ophthalmopathy Quality of Life Scale | month 1，month 3，month 6
  The Graves' Ophthalmopathy Quality of Life (GO-QOL) questionnaire [4]includes visual functioning and psychosocial functioning. A raw score of each part is calculated by adding each score of 8 question, namely 1, 2, or 3 for each question which means marked, mild, or absent limitation, the final score ranging from 0 (full limitation) to 100 (no limitation) is calculated as the following rule: (raw score - 8) ÷ 16 × 100]. GO-QOL will be completed at screening, week 0, week 4 and week 12. The data will also be recorded to assess activity of TAO and impact on quality of life respectively.
  The GO-QOL is a 16-item self-administered questionnaire used to assess the perceived effects of TAO by the patients on their daily physical and psychosocial functioning.
inflammatory markers changes | month 1，month 3，month 6
  Serum inflammatory markers （systemic）including neutrophil, lymphocyte, platelet, monocyte, WBC, NLR, PLR, MLR, SII,SIRI, PIV, WMR and others.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Liang, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No